CLINICAL TRIAL: NCT07113795
Title: Clinical Study on the Integration of Traditional Chinese Medicine Xu Gua Therapy With Mesenchymal Stem Cells for the Treatment of Crohn's Disease-Associated Anal Fistula.
Brief Title: Clinical Study on the Integration of Traditional Chinese Medicine Virtual Hanging Therapy With Mesenchymal Stem Cells for the Treatment of Crohn's Disease-Associated Anal Fistula.
Acronym: VH-MSC-CDAF
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Anorectal Center of Nanjing Hospital of Traditional Chinese Medicine (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BE2022674
Record Dates: First submitted 2025-05-19; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease With Perianal Fistulas
Keywords: Traditional Chinese Medicine; Virtual Hanging therapy; Mesenchymal Stem Cells; Crohn's Disease-Associated Anal Fistula; Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Association Group (Experimental): receiving a combination of TCM dummy therapy and mesenchymal stem cell injection therapy
  Interventions: Procedure: TCM dummy therapy combined with mesenchymal stem cell injection therapy
- Dummy Line Therapy Group (Active Comparator): treated solely with dummy line therapy
  Interventions: Procedure: Dummy Line Therapy Group
- MSC Group (Active Comparator): administered only mesenchymal stem cell injection therapy
  Interventions: Procedure: MSC Group

INTERVENTIONS:
Procedure: TCM dummy therapy combined with mesenchymal stem cell injection therapy — Combines TCM dummy therapy with mesenchymal stem cell injection, integrating traditional local stimulation and modern stem cell regenerative mechanisms.
  Arms: Association Group
Procedure: Dummy Line Therapy Group — Utilizes traditional thread-embedding techniques, placing specialized threads at specific sites to effectively drain inflammatory exudates and necrotic materials.
  Arms: Dummy Line Therapy Group
Procedure: MSC Group — Administers mesenchymal stem cell injections directly to target areas, leveraging their differentiation and anti-inflammatory properties to enhance tissue repair.
  Arms: MSC Group

SUMMARY:
To evaluate the efficacy and safety of TCM virtual hanging therapy combined with mesenchymal stem cellsin the treatment of CD anal fistula. To establish the standard of clinical diagnosis and treatment and thestandard procedure of operation for the treatment of CD anal fistula by virtual hanging therapy combinedwith mesenchymal stem cells.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent form.

Diagnosis of Crohn's disease (CD) confirmed at least 6 months prior to screening, based on the Chinese Consensus on Diagnosis and Treatment of Inflammatory Bowel Disease (2018, Beijing).

Crohn's Disease Activity Index (CDAI) score ≤220, indicating inactive or mildly active CD.

Presence of complex anal fistula confirmed by clinical and MRI evaluation.

Age 18-60 years (inclusive), regardless of sex.

Negative serum/urine pregnancy test for women of childbearing potential; all participants must agree to use effective contraception during and for 6 months after the trial.

Good general health status confirmed by medical history and relevant examinations.

Exclusion Criteria:

CDAI >220 or requiring immediate treatment for active CD.

Patients with rectal/anal stenosis or active proctitis (due to procedural limitations).

Presence of abscess >2 cm unless treated ≥2 weeks prior to the trial.

History of fistula surgery (except drainage or seton placement), concurrent need for perianal surgery unrelated to fistula, or anticipated need for such surgery within 24 weeks post-treatment.

Systemic steroid therapy within 4 weeks prior to screening.

Abnormal laboratory results:

Liver function: Total bilirubin ≥1.5×ULN; aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥2.5×ULN.

Renal function: Creatinine clearance <60 mL/min or serum creatinine ≥1.5×ULN (measured or calculated by Cockcroft-Gault formula).

Current or history of malignancy (including fistula-related carcinoma).

Severe, progressive, or uncontrolled hepatic, hematologic, gastrointestinal (excluding CD), endocrine, pulmonary, cardiac, neurologic, psychiatric, or cerebral diseases.

HIV/syphilis antibody positivity, active HCV/HBV infection, or active tuberculosis.

Known allergy to antibiotics or trial-related agents (e.g., penicillin, streptomycin, gentamicin, aminoglycosides, human serum albumin, human platelet lysate, DMEM cell culture medium, or bovine-derived materials).

Intolerance to anesthesia or contraindications to MRI scanning (e.g., pacemaker, hip prosthesis, severe claustrophobia, gadolinium allergy).

Pregnancy, lactation, or refusal to use effective contraception during and for 6 months post-trial.

Major surgery or severe trauma within the past 6 months.

History of alcohol/drug abuse within 6 months prior to enrollment.

Use of investigational drugs within 12 weeks (84 days) prior to screening.

Inability to comply with the study protocol or other conditions deemed unsuitable by investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
CD anal fistula healing rate | From enrollment to the end of treatment at 24 weeks
  Post-treatment healing rate of Crohn's disease-related anal fistula, defined as clinical closure of all external fistula openings in patients, combined with MRI-confirmed fistula tract healing.

SECONDARY OUTCOMES:
CDAI | From enrollment to the end of treatment at 24 weeks
  A clinical scoring system to quantify disease activity in Crohn's disease (CD) patients, integrating symptoms (e.g., abdominal pain, diarrhea) and laboratory parameters (e.g., hemoglobin, ESR).0~600(~600, theoretically no upper limit).Higher scores indicate worse disease activity (poorer outcome).
PDAI | From enrollment to the end of treatment at 24 weeks
  A standardized tool to assess the severity of perianal complications (e.g., fistulas, abscesses) in Crohn's disease, combining clinical symptoms (e.g., pain, discharge) and imaging findings.0-20.Higher scores indicate worse perianal disease activity (poorer outcome).
IBDQ | From enrollment to the end of treatment at 24 weeks
  A validated patient-reported outcome measure evaluating the quality of life in IBD patients across physical, emotional, and social domains.32-224.Higher scores indicate better health-related quality of life (better outcome).
Van Assche | From enrollment to the end of treatment at 24 weeks
  An MRI-based scoring system for perianal fistulas, grading anatomical complexity (e.g., fistula branches, abscesses) and inflammatory activity to guide therapeutic strategies.0-12.Higher scores indicate more severe perianal fistulizing disease on MRI (poorer outcome).
VAS | From enrollment to the end of treatment at 24 weeks
  A unidimensional pain assessment tool where patients mark their pain intensity on a 10-cm line (0=no pain, 10=worst pain).
Wexner | From enrollment to the end of treatment at 24 weeks
  A validated scoring system to evaluate constipation severity based on stool frequency, straining, incomplete evacuation, and associated symptoms (e.g., abdominal bloating).0-20.Higher scores indicate worse fecal incontinence severity (poorer outcome).
Erythrocyte Sedimentation Rate (ESR) | From enrollment to the end of treatment at 24 weeks
  A nonspecific inflammatory marker reflecting the rate at which red blood cells settle in a tube over one hour; elevated in infections, autoimmune diseases, or chronic inflammation.
Fecal Calprotectin | From enrollment to the end of treatment at 24 weeks
  A stool biomarker of intestinal inflammation, reflecting neutrophil activity; used to differentiate inflammatory bowel disease (IBD) from functional gastrointestinal disorders.
C-reactive Protein (CRP) | From enrollment to the end of treatment at 24 weeks
  An acute-phase protein synthesized by the liver; elevated serum levels indicate systemic inflammation, infection, or tissue damage.
Anorectal Manometry | From enrollment to the end of treatment at 24 weeks
  Primary outcome measures: Anal Resting Pressure (basal sphincter pressure at rest; normal 40-80mmHg; <40mmHg=incontinence risk), Maximum Anal Squeeze Pressure (peak voluntary squeeze; normal 100-200mmHg; <100mmHg=sphincter impairment), Recto-anal Pressure Gradient (rectal-anal pressure difference; normal -20 to -50mmHg; positive=dyssynergic defecation). Secondary: First Sensation Volume (minimal rectal balloon volume for sensation; normal 10-30mL; >30mL=hyposensitivity), Urge Volume (volume for sustained defecation urge; normal 40-80mL; >80mL=severe sensory dysfunction), Max Rectal Volume (max tolerated distension; normal 120-200mL; <120mL=low compliance), Balloon Expulsion Time (time to expel 50mL balloon; normal ≤60s; >60s=pelvic dyssynergia), Anal High Pressure Zone Length (axial sphincter length; normal 2.0-4.0cm; <2.0cm=anatomical defect).

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Hospital of Traditional Chinese Medicine (Affiliated Hospital of Nanjing University of Chinese Medicine), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
This is a single-center study without involvement of other institutions.